CLINICAL TRIAL: NCT00639899
Title: Selective Retrograde Venography and Sclerotherapy of Internal Spermatic Veins and Associated Venous Bypasses and Retro-Peritoneal Collateral in Patients With Varicocele and Hypertrophy of Prostate
Brief Title: The Effect of Spermatic Vein Embolization on Prostatic Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maaynei Hayesha Medical Center (Other)
Responsible Party: Dr Uriel Levinger, Maaynei Hayesha Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVS-001-IL
Record Dates: First submitted 2008-03-09; First posted 2008-03-20 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Varicocele
Keywords: Varicocele
MeSH Terms: conditions — Varicocele | interventions — Sclerotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sclerotherapy — Super-selective retrograde venography and sclerotherapy of internal spermatic veins and associated venous bypasses and retro-peritoneal collateral

SUMMARY:
In varicocele the venous pressure in the prostatic bed is increased .This may result in raised hydrostatic pressure which in turn may stimulate prostatic hypertrophy.

Restoring normal venous drainage is expected to lower hydrostatic pressure followed by inhibition of prostatic growth and possibly leading regression in prostatic dimensions.

DETAILED DESCRIPTION:
35 male patients, aged 45 years or older, with documented benign prostatic hypertrophy (BPH)and varicocele as visualized by ultrasound and/or termography examination will be enrolled.

Each patient will undergo a full urologic examination to exclude possible malignancy as well as a thorough medical examination to establish eligibility for treatment.

In all selected patients the varicocele will be obliterated by means of embolization of the spermatic veins.

The patients will be followed every three months by abdominal ultrasound as well as by serial PSA for a period of 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age > 45 < 80 years
* BPH
* Bilateral varicocele.

Exclusion Criteria:

* Coagulation disturbance
* CHF
* Malignancy
* Renal failure.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety performance of the procedure. Reduction of above 20% in prostatic calculated volume. | 1 year

SECONDARY OUTCOMES:
Reduction of above 20% in nocturia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Levinger, MD, Principal Investigator — Maaynei Hayeshua Medical Center
Locations (1):
- Maaynei Hayeshua Medical Center, Bnei Brak, Israel